CLINICAL TRIAL: NCT01973244
Title: A Randomised, Open-labelled, Active-controlled, Multinational, Dose-escalation Trial Investigating Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of a Single Dose of Long-acting Growth Hormone (NNC0195-0092, Somapacitan) Compared to Daily Dosing of Norditropin® SimpleXx® in Children With Growth Hormone Deficiency
Brief Title: A Trial Investigating Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of a Single Dose of Long-acting Growth Hormone (Somapacitan) Compared to Daily Dosing of Norditropin® SimpleXx® in Children With Growth Hormone Deficiency
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN8640-4042; 2013-000013-20 (EudraCT Number); U1111-1138-2206 (Other: WHO); REec-2014-0688 (Registry Identifier: Spanish Register of Clinical Studies (REec)); JapicCTI-142663 (Registry Identifier: JAPIC)
Record Dates: First submitted 2013-10-22; First posted 2013-10-31 (Estimated); Last update posted 2020-12-24 (Actual); Status verified 2020-12

CONDITIONS: Growth Hormone Disorder; Growth Hormone Deficiency in Children
MeSH Terms: interventions — somapacitan; NNC0195-0092; Human Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- NNC0195-0092 (somapacitan) (Experimental)
  Interventions: Drug: somapacitan
- Norditropin® (Active Comparator)
  Interventions: Drug: somatropin

INTERVENTIONS:
Drug: somapacitan — A single dose administered subcutaneously (s.c., under the skin) of 4 different doses of NNC0195-0092 in an escalating order.
  Each subject will be allocated to one dose level only. After completion of each dose cohort, a safety evaluation will be conducted prior to dose escalation.
  Other Names: NNC0195-0092
  Arms: NNC0195-0092 (somapacitan)
Drug: somatropin — Administered subcutaneously (s.c., under the skin) once daily for 7 days. The daily dose is 0.03 mg/kg/day.
  Arms: Norditropin®

SUMMARY:
This trial is conducted in Europe and Asia. The aim of the trial is to investigate safety, tolerability, pharmacokinetics (the exposure of the trial drug in the body) and pharmacodynamics (the effect of the investigated drug on the body) of a single dose of long-acting growth hormone (NNC0195-0092, somapacitan) compared to daily dosing of Norditropin® SimpleXx® (somatropin) in children with growth hormone deficiency.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of GHD (growth hormone deficiency) as defined by two different GH (growth hormone) stimulation tests, peak GH level below or equal to 7.0 ng/ml. For children with three or more pituitary hormone deficiencies only one GH stimulation test will be needed. If in accordance with country specific practice, growth hormone deficiency can be defined by only one GH stimulation test, peak GH level below or equal to 7.0 ng/ml.
* Pre-pubertal children at screening. Boys: Tanner stage 1 and age above or equal to 6 years and below 13 years. Girls: Tanner stage 1 and age above or equal to 6 years and below 12 years
* Body weight above or equal to 16.0 kg and below or equal to 50.0 kg
* Stable GH replacement treatment for at least 3 months

Exclusion Criteria:

* History or presence of malignancy
* Overt diabetes mellitus (fasting blood glucose above or equal to 7.0 mmol/l)

Ages: 6 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2013-12-16 (Actual); Primary Completion 2014-11-04 (Actual); Study Completion 2014-11-04 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) | From first administration of trial product and up until day 35 (final visit)

SECONDARY OUTCOMES:
The area under the insulin-like growth factor I (IGF-I) concentration-time curve | From 0 to 168 hours after dosing

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (21):
- Austria (3):
  - Novo Nordisk Investigational Site, Graz
  - Novo Nordisk Investigational Site, Linz
  - Novo Nordisk Investigational Site, Vienna
- Novo Nordisk Investigational Site, Brussels, Belgium
- France (2):
  - Novo Nordisk Investigational Site, Paris
  - Novo Nordisk Investigational Site, Toulouse
- Israel (5):
  - Novo Nordisk Investigational Site, Haifa
  - Novo Nordisk Investigational Site, Jerusalem
  - Novo Nordisk Investigational Site, Kfar Saba
  - Novo Nordisk Investigational Site, Petah Tikva
  - Novo Nordisk Investigational Site, Tel Litwinsky
- Novo Nordisk Investigational Site, Skopje, North Macedonia
- Novo Nordisk Investigational Site, Bergen, Norway
- Novo Nordisk Investigational Site, Ljubljana, Slovenia
- Spain (4):
  - Novo Nordisk Investigational Site, Barcelona
  - Novo Nordisk Investigational Site, Esplugues Llobregat(Barcelona)
  - Novo Nordisk Investigational Site, Santiago de Compostela
  - Novo Nordisk Investigational Site, Vitoria-Gasteiz
- Novo Nordisk Investigational Site, Stockholm, Sweden
- Switzerland (2):
  - Novo Nordisk Investigational Site, Basel
  - Novo Nordisk Investigational Site, Geneva

REFERENCES:
- [Background] Juul Kildemoes R, Hojby Rasmussen M, Agerso H, Overgaard RV. Optimal Monitoring of Weekly IGF-I Levels During Growth Hormone Therapy With Once-Weekly Somapacitan. J Clin Endocrinol Metab. 2021 Jan 23;106(2):567-576. doi: 10.1210/clinem/dgaa775. PMID 33313798
- [Derived] Papathanasiou T, Agerso H, Damholt BB, Hojby Rasmussen M, Kildemoes RJ. Population Pharmacokinetics and Pharmacodynamics of Once-Daily Growth Hormone Norditropin(R) in Children and Adults. Clin Pharmacokinet. 2021 Sep;60(9):1217-1226. doi: 10.1007/s40262-021-01011-3. Epub 2021 Apr 17. PMID 33864240
- [Derived] Juul RV, Rasmussen MH, Agerso H, Overgaard RV. Pharmacokinetics and Pharmacodynamics of Once-Weekly Somapacitan in Children and Adults: Supporting Dosing Rationales with a Model-Based Analysis of Three Phase I Trials. Clin Pharmacokinet. 2019 Jan;58(1):63-75. doi: 10.1007/s40262-018-0662-5. PMID 29671202
- [Derived] Battelino T, Rasmussen MH, De Schepper J, Zuckerman-Levin N, Gucev Z, Savendahl L; NN8640-4042 Study Group. Somapacitan, a once-weekly reversible albumin-binding GH derivative, in children with GH deficiency: A randomized dose-escalation trial. Clin Endocrinol (Oxf). 2017 Oct;87(4):350-358. doi: 10.1111/cen.13409. Epub 2017 Aug 8. PMID 28656605
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com